CLINICAL TRIAL: NCT06986655
Title: The Effect of an Augmented Reality Game on Pain, Fear, and Care Satisfaction Levels During Allergy Testing in Children Aged 4-12 Years: A Randomized Controlled Trial
Brief Title: The Effect of an Augmented Reality Game on Pain, Fear, and Care Satisfaction Levels During Allergy Testing in Children Aged 4-12 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Collaborators: Koç University Hospital (Unknown)
Responsible Party: Principal Investigator, Enes Simsek, Principal Investigator, Koç University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2023.206.IRB1.068
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Augmented Reality
Keywords: allergy; pediatric; augmented reality; pain; anxiety; care satisfaction
MeSH Terms: conditions — Hypersensitivity; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (AR Group) (Experimental): Children in this group will be exposed to an augmented reality game during the allergy testing procedure. The game will be used as a distraction method to potentially reduce pain and fear, and enhance care satisfaction.
  Interventions: Other: Augmented Reality
- Control Arm (Standard Care Group) (No Intervention): Children in this group will undergo allergy testing following standard clinical procedures without any AR intervention or distraction.

INTERVENTIONS:
Other: Augmented Reality — In this intervention children will play an augmented reality game during the allergy testing procedure. The game will be used as a distraction method to potentially reduce pain and fear, and enhance care satisfaction.
  Arms: Intervention Arm (AR Group)

SUMMARY:
The aim of this study is to examine the effects of augmented reality (AR) games on pain, fear, and care satisfaction, and to contribute to the literature on innovative interventions that enhance the healthcare experiences of children undergoing allergy testing.

H1: The pain level of children undergoing allergy testing in the AR group is lower than that of children in the control group.

H2: The fear level of children undergoing allergy testing in the AR group is lower than that of children in the control group.

H3: The care satisfaction level of children undergoing allergy testing in the AR group is higher than that of children in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 4 and 12 years.
* Scheduled to undergo an allergy test.
* No visual impairments that would interfere with the use of augmented reality -applications.
* No use of anxiolytic or analgesic medications within the last six hours.
* Willing to participate in the study, with parental/legal guardian consent as applicable.

Exclusion Criteria:

* Younger than 4 years or older than 12 years.
* Not scheduled for an allergy test.
* Presence of visual impairments.
* Use of anxiolytic or analgesic medications within the last six hours.
* Unwilling to participate in the study or lacking informed consent.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Pain Level | Immediately after the allergy testing procedure.
  Wong-Baker FACES Pain Rating Scale is used for this measurement. This scale consists of six facial expressions that represent increasing levels of pain, ranging from "No pain" (0 points) to "Worst pain" (10 points). Children are asked to point to the face that best matches the pain they are experiencing.
Fear level | Immediately before and after the allergy testing procedure.
  Children's Fear Scale is used for the fear measurement. This self-report tool consists of six facial expressions corresponding to fear levels, rated from 0 (no fear) to 10 (maximum fear), in increments of two points. Children are asked to select the face that best represents their emotional state.
Care Satisfaction | Immediately after the allergy testing procedure.
  Visual Analog Scale (VAS) for Care Satisfaction is used to assess the child's satisfaction with the care received during the allergy test. The score ranges from 0 ("Not satisfied at all") to 10 ("Completely satisfied").

CONTACTS AND LOCATIONS:
Overall Officials: Remziye Semerci Şahin, Assistant professor, Study Director — Koç University
Locations (1):
- Koç University Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No